CLINICAL TRIAL: NCT01592500
Title: Safety and Dose Finding Study of Different MOD-4023 Dose Levels Compared to Daily r-hGH Therapy in Pre-pubertal Growth Hormone Deficient Children
Brief Title: Safety and Efficacy Phase 2 Study of Long-acting hGH (MOD-4023) in Growth Hormone Deficient Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-4-004; 2011-004553-60 (EudraCT Number)
Record Dates: First submitted 2012-05-02; First posted 2012-05-07 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Pediatric Growth Hormone Deficiency
Keywords: GHD; r-hGH; Long-acting
MeSH Terms: interventions — MOD-4023; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MOD-4023 low dose (Experimental): Once weekly subcutaneous injection of long acting r-hGH (MOD-4023)
  Interventions: Drug: MOD-4023
- MOD-4023 middle dose (Experimental): Once weekly subcutaneous injection of long acting r-hGH (MOD-4023)
  Interventions: Drug: MOD-4023
- MOD-4023 high dose (Experimental): Once weekly subcutaneous injection of long acting r-hGH (MOD-4023)
  Interventions: Drug: MOD-4023
- Genotropin (Active Comparator): Once daily subcutaneous injection of Somatropin (r-hGH; Genotropin)
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: MOD-4023 — Once weekly subcutaneous injection
  Arms: MOD-4023 high dose; MOD-4023 low dose; MOD-4023 middle dose
Drug: Somatropin — Once daily subcutaneous injection of Genotropin
  Other Names: Genotropin
  Arms: Genotropin

SUMMARY:
This is a phase II, open label, active-controlled, randomized safety and dose finding study of different MOD-4023 dose levels compared to daily r-hGH therapy in pre-pubertal growth hormone deficient children.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-pubertal child aged ≥ 3 yrs old and not above 10 years for girls or 11 years for boys with either isolated GHD, or GH insufficiency as part of multiple pituitary hormone deficiency.
2. Confirmed diagnosis of GHD by two different GH provocation tests defined as a peak plasma GH level of ≤7 ng/ml, determined by central laboratory using a validated assay .
3. Bone age (BA) is not older than chronological age and should be no greater than 9 years for girls and 10 years for boys.
4. Without prior exposure to any r-hGH therapy.
5. Normal birth size, birth weight and length for gestational age
6. Impaired height and height velocity defined as:

   1. Height (HT) of at least 2.0 standard deviations (SD) below the mean height for chronological age (CA) and gender according to the standards from Prader et. al, 1989 , (HT SDS ≤ -2.0).
   2. Annualized height velocity (HV) below the 25th percentile for CA (HV <-0.7 SDS) and gender according to the standards of Prader et al (1989). The interval between two height measurements should be at least 6 months before inclusion.
7. BMI must be within ±2 SD of mean BMI for the chronological age and sex according to the 2000 CDC standards.
8. Baseline IGF-I level of at least 1 SD below the mean IGF-I level standardized for age and sex (IGF-I SDS ≤ -1.0) according to the central laboratory reference values;
9. 12. Written informed consent of the parent or legal guardian of the patient and assent of the patient (if the patient can read).

Exclusion Criteria:

1. Children with past or present intracranial tumor growth as confirmed by an MRI scan (with contrast).
2. History of radiation therapy or chemotherapy.
3. Malnourished children defined as:

   1. Serum albumin below the lower limit of normal (LLN) according to the reference ranges of central laboratory;
   2. Serum iron below the lower limit of normal (LLN) according to the reference ranges of central laboratory;
   3. BMI < -2 SD for age and sex;
4. Children with psychosocial dwarfism.
5. Children born small for gestational age (SGA - birth weight and/or birth length < -2 SD for gestational age).
6. Presence of anti-hGH antibodies at screening.
7. Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to, chronic diseases like renal insufficiency, spinal cord irradiation, etc.
8. Patients with diabetes mellitus.
9. Patients with impaired fasting sugar (based on WHO; fasting blood sugar >110 mg/dl or 6.1 mmol/l) after repeated blood analysis.
10. Chromosomal abnormalities and medical "syndromes" (Turner's syndrome, Laron syndrome, Noonan syndrome, Prader-Willi Syndrome, Russell-Silver Syndrome, SHOX mutations/deletions and skeletal dysplasias), with the exception of septo-optic dysplasia.
11. Closed epiphyses.
12. Concomitant administration of other treatments that may have an effect on growth such as anabolic steroids and methylphenidate for attention deficit hyperactivity disorder (ADHD), with the exception of hormone replacement therapies (thyroxine, hydrocortisone, desmopressin (DDAVP))
13. Children requiring glucocorticoid therapy (e.g. asthma) who are taking a dose of greater than 400 µg/d of inhaled budesonide or equivalents for longer than 1 month during a calendar year.
14. Major medical conditions and/or presence of contraindication to r-hGH treatment.
15. Known or suspected HIV-positive patient, or patient with advanced diseases such as AIDS or tuberculosis.
16. Drug, substance, or alcohol abuse.
17. Known hypersensitivity to the components of study medication.
18. Other causes of short stature such as coeliac disease, hypothyroidism and rickets.
19. The patient and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct.
20. Participation in any other trial of an investigational agent within 30 days prior to Screening.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2012-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Zadik, MD, Principal Investigator — Kaplan Medical Center, Israel
Locations (4):
- Children's Hospital "P. A. Kyriakou", Athens, Greece
- Hungary (2):
  - Buda Children's Hospital, Budapest
  - Heim Pal Children's Hospital, Budapest
- Children's University Hospital, Košice, Slovakia

REFERENCES:
- [Derived] Zelinska N, Iotova V, Skorodok J, Malievsky O, Peterkova V, Samsonova L, Rosenfeld RG, Zadik Z, Jaron-Mendelson M, Koren R, Amitzi L, Raduk D, Hershkovitz O, Hart G. Long-Acting C-Terminal Peptide-Modified hGH (MOD-4023): Results of a Safety and Dose-Finding Study in GHD Children. J Clin Endocrinol Metab. 2017 May 1;102(5):1578-1587. doi: 10.1210/jc.2016-3547. PMID 28323965

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin
Started | 14 (Randomized Participants) | 15 | 14 | 13 (Randomized Participants)
Completed | 13 | 15 | 14 | 11
Not Completed | 1 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin | Total
Number analyzed (Participants) | 13 | 15 | 14 | 11 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 15 | 14 | 11 | 53
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 5 | 3 | 17
  Male | 10 | 9 | 9 | 8 | 36

OUTCOME MEASURES:

1. Primary Outcome: Annual Height Velocity
Description: Annual Height Velocity in cm/year measured after 12 months of treatment
Time Frame: 12 months of treatment
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin
Number analyzed (Participants) | 13 | 15 | 13 | 11
cm/year | 10.4 (2.6) | 11.0 (2.3) | 11.9 (3.5) | 12.5 (2.1)

2. Secondary Outcome: Height Velocity at 6 Months
Description: Annualized Height Velocity in cm/year measured after 6 months of treatment
Time Frame: After 6 months of treatment
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin
Number analyzed (Participants) | 13 | 15 | 13 | 11
cm/year | 11.8 (3.6) | 12.5 (2.4) | 13.5 (5.0) | 15.0 (2.9)

3. Secondary Outcome: Change in Height Standard Deviation Score (SDS)
Description: Change in height standard deviation score from baseline (compared to normal population of same age group and sex). Height SDS was calculated as height minus reference mean height divided by SD of the reference mean height
Time Frame: After 6 and 12 months of treatment
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin
Number analyzed (Participants) | 13 | 15 | 13 | 11
score on a scale
  After 6 months of treatment | 0.65 (0.36) | 0.75 (0.25) | 0.90 (0.39) | 1.00 (0.35)
  After 12 months of treatment | 1.09 (0.53) | 1.19 (0.49) | 1.45 (0.61) | 1.51 (0.47)

4. Secondary Outcome: Change in IGF-1 Standard Deviation Score
Description: Change in IGF-1 standard deviation score from reference population mean of same age group and sex (WHO source). IGF-1 SDS was calculated as IGF-1 result minus reference mean IGF-1 result divided by SD of the reference mean IGF-1 value.
Time Frame: Once monthly on day 4 after the last dose
Population: No data were scheduled to be collected for Week 23 in the Genotropin Arm/Group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin
Number analyzed (Participants) | 13 | 15 | 14 | 11
score on a scale
  Week 1 | -1.86 (0.817) | -1.94 (0.899) | -2.13 (0.887) | -2.12 (0.813)
  Week 10 | -1.03 (0.902) | -0.279 (0.891) | -0.001 (1.164) | -0.515 (1.238)
  Week 14 | -1.07 (0.553) | -0.275 (0.772) | -0.058 (1.067) | -0.557 (1.216)
  Week 18 | -0.815 (0.733) | 0.189 (0.707) | -0.083 (1.299) | -0.310 (0.896)
  Week 22 | -0.958 (0.673) | -0.188 (0.684) | 0.023 (0.964) | -0.495 (1.108)
  Week 23: number analyzed (Participants) | 13 | 15 | 14 | 0
  Week 23 | -1.70 (0.741) | -1.48 (0.653) | -1.47 (0.865) |
  Week 26 | -0.725 (0.801) | 0.088 (0.803) | -0.011 (1.084) | -0.235 (0.919)
  Month 9 | -0.119 (0.921) | 0.184 (0.905) | 0.261 (1.108) | 0.124 (1.071)
  Month 12 | -0.458 (1.194) | -0.029 (1.296) | 0.358 (0.709) | -0.015 (1.485)

ADVERSE EVENTS:
Arm/Group | MOD-4023 Low Dose | MOD-4023 Middle Dose | MOD-4023 High Dose | Genotropin
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/14 | 0/11
Other Adverse Events (participants affected / at risk) | 10/13 | 10/15 | 10/14 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOD-4023 Low Dose (N=13) | MOD-4023 Middle Dose (N=15) | MOD-4023 High Dose (N=14) | Genotropin (N=11)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 3 | 1
Iron Deficiency Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 1 | 1
Secondary Adrenocortical Insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Amblyopia (Eye disorders) | 1 | 0 | 0 | 0
Astigmatism (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Eye Inflammation (Eye disorders) | 1 | 0 | 0 | 0
Eyelid Oedema (Eye disorders) | 1 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Acetonaemic Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 1
Chest Pain (General disorders) | 1 | 0 | 0 | 0
Injection Site Erythema (General disorders) | 1 | 0 | 1 | 0
Injection Site Haematoma (General disorders) | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 0 | 1 | 0
Injection Site Pruritus (General disorders) | 0 | 0 | 1 | 0
Injection Site Swelling (General disorders) | 1 | 0 | 1 | 0
Edema Peripheral (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Sphincter of Oddi Dysfunction (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 2
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Helminthic Infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 2
Pulpitis Dental (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 2 | 3
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 2 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 2 | 0
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus Cyst (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Body Temperature Increased (Investigations) | 1 | 0 | 0 | 0
Hemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0
Insulin-Like Growth Factor Increased (Investigations) | 0 | 0 | 1 | 0
Red Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 1
Thyroxine Decreased (Investigations) | 0 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 0 | 1
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes